CLINICAL TRIAL: NCT04270851
Title: Colorectal Liver Metastases: Novel Assessment Tools for Technical Resectability (The CoNoR Study)
Brief Title: Colorectal Liver Metastases: Novel Assessment Tools for Technical Resectability
Acronym: CoNoR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Manchester (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government); Perspectum (Industry); The Christie NHS Foundation Trust (Other); The Royal College of Surgeons of England (Other)
Responsible Party: Principal Investigator, Kat Parmar, Clinical Research Fellow, University of Manchester
Other Study IDs: IRAS ID 266961
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Cancer; Cancer Metastatic; Colorectal Cancer; Liver Metastasis Colon Cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Borderline Resectability: Patients with colorectal liver metastases where the decision-making on technical resectability is difficult, i.e. 'borderline resectable,' where a group of liver surgeons might reasonably be expected to find the decision whether to operate to be challenging. A group of up to 20 such patients will undergo pre-operative LiMAx test and HepaT1ca pre-operative scanning. Recruited participants' data will be used to create anonymised online case scenarios to be used in a survey, assessing whether liver surgeons find these pre-operative assessments helpful in their decision-making on technical resectability.
  Interventions: Diagnostic Test: LiMAx test; Diagnostic Test: HepaT1ca magnetic resonance scan

INTERVENTIONS:
Diagnostic Test: LiMAx test — The LiMAx test is a fully licenced liver function test, testing liver maximum capacity via a breath test.
Diagnostic Test: HepaT1ca magnetic resonance scan — The HepaT1ca scan is a pre-operative magnetic resonance scan providing a detailed report permitting interactive virtual pre-operative planning prior to liver surgery.

SUMMARY:
The CoNoR study aims to assess whether the use of the LiMAx test and the HepaT1ca pre-operative planning magnetic resonance scan impact upon technical resectability decision-making in colorectal liver metastases (CLM).

DETAILED DESCRIPTION:
The CoNoR Study will occur via 4 workstreams:

1. Systematic review of all published criteria for colorectal liver metastases (CLM) technical resectability (systematic review protocol published on PROSPERO database: https://www.crd.york.ac.uk/prospero/display_record.php?RecordID=136748
2. Expert interviews: Interviews with liver surgeons and radiologists to assess current standard practice in CLM technical resectability decision-making and role for novel assessment tools
3. Online questionnaire: Online international questionnaire of liver surgeons to assess current standard practice in CLM technical resectability decision-making and role for novel assessment tools, in additional to identifying clinical scenarios in which these tools may be of greatest benefit
4. Online case-based survey: Recruitment of 10-20 participants with 'difficult decisions' regarding technical resectability, and consent to use results from pre-operative assessments to create anonymised online case-based survey. Participants will consent to have two additional pre-operative assessments: the LiMAx tests and the HepaT1ca magnetic resonance scan. These results from these additional tests will also be used in the online survey, We will recruit international liver surgeons to complete this online survey, where they will be asked to provide an opinion on technical resectability for each individual case scenario, and to specify their operative plan, both before and after seeing the results of these novel assessment tools. We will assess for change in decision-making on resectability, and change in operative plan after seeing these test results. We will also assess for level of agreement between liver surgeons on each scenario, and identify where they difficult decisions persist.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 16 years of age with histologically verified adenocarcinoma of the colon or rectum and radiological evidence of liver metastases
2. Discussion at regional hepatobiliary multidisciplinary team meeting
3. Hepatobiliary surgical opinion that their case represents a potentially difficult decision regarding technical resectability
4. Ability to provide written informed consent

Exclusion Criteria:

1. Presence of a medical or psychiatric condition impairing the ability to give informed consent
2. Presence of any other serious uncontrolled medical condition
3. Patients under 16 years old
4. Contra-indications to magnetic resonance scanning

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically verified adenocarcinoma of the colon or rectum and radiological evidence of liver metastases
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Change in decision making on technical resectability | One year
  Liver surgeons will view the standard pre-operative assessment results and decide if each case scenario is 'technically resectable.' They will then view the results from these two additional pre-operative tests (LiMAx and HepaT1ca), and decide again. We will measure for any change in decision making after viewing the novel test results.

SECONDARY OUTCOMES:
Change in operative plan | One Year
  Liver surgeons will view the standard pre-operative assessment results and specify their operative plan for each clinical scenario. They will then view the results from these two additional pre-operative tests (LiMAx and HepaT1ca), and specify their operative plan again. We will measure for any change in decision making in their operative plan after viewing the novel test results.
Level of agreement between liver surgeons on technical resectability | One Year
  For all participating surgeons, we will measure the level of agreement between them when they decide if each case scenario is technically resectable.

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parmar KL, O'Reilly D, Valle J, Braun M, Malcomson L, Jones RP, Balaa F, Rees M, Welsh FKS, Filobbos R, Renehan AG. Protocol for the CoNoR Study: A prospective multi-step study of the potential added benefit of two novel assessment tools in colorectal liver metastases technical resectability decision-making. BMJ Open. 2023 Mar 30;13(3):e059369. doi: 10.1136/bmjopen-2021-059369. PMID 36997247